CLINICAL TRIAL: NCT06069674
Title: Use of Cerebral Biomarkers in Minor Traumatic Brain Injury in the Emergency Unit
Acronym: CerBio-mTBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, COVINO MARCELLO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5571
Record Dates: First submitted 2023-05-19; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Brain Injuries, Traumatic; Trauma; Trauma, Nervous System
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Trauma, Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum dosage of GFAP and UCH-L1 — blood test execution as per usual care in the ED

SUMMARY:
The use of serum biomarkers in the setting of the emergency department (ED) has been well characterized over the years as an adjunctive tool for the clinician in the setting of complex decision making. In this regard, the serum dosage of glial fibrillary acidic protein (GFAP) and ubiquitin C-terminal hydrolase L1 (UCH-L1) has been evaluated in a series of successful multicenter prospective studies as a potentially useful marker of, respectively, glial and neuronal damage in the setting of mild traumatic brain injury (mTBI), which is defined as a brain injury (concussion) secondary to trauma with a GCS (Glasgow coma scale) score of 13-15. It seems that both markers are detectable in serum less than 1 hour after the traumatic event, with highest levels appearing at around 2 hours, and are capable of distinguishing between patients with traumatic brain injury from those without acute brain injury after trauma. Furthermore, they seem to possess a high negative predictive value for detection of intracranial injuries at head CT-scan as well as the need of neurosurgical intervention after head trauma.

Mild traumatic brain injury is one of the most frequent chief-complaints for patients presenting to emergency departments worldwide. At present, head CT scan is the gold standard diagnostic test for the identification of potentially life-threatening intra-cranial injuries. Although effective in the identification of serious lesions which might require neurosurgical intervention or in-hospital prolonged observation, the extensive use of head CT scan in mTBI has been questioned due to the potential risks related to radiation exposure, as well as unnecessary deployment of ED resources and increased costs, considering that the prevalence of CT-detected intra-cranial injury in mTBI is around 5-10%.

For this reason, a number of international clinical guidelines suggest several Clinical Decision Rules (CDR) and algorithms to guide the clinician in the correct management of these patients, in particular in the difficult feat of identifying those patients who don't need to perform neuroradiological evaluation (CT scan or MRI) in the setting of the ED, without the risk to overlook potentially fatal brain injuries.

The adjunctive role of these biomarkers has been well characterized in the setting of mTBI. It seems they correlate well with neurological damage as well as with the presence of CT abnormalities, and it seems that they might perform better than clinical evaluation alone.

Nonetheless, according to current international guidelines and several systematic reviews and meta-analysis, patients who present with mTBI and risk factors for bleeding and delayed bleeding (such as known coagulopathy, patients on blood thinners or advanced age), need to perform CT scan plus clinical observation or even serial CT scans when the risk of delayed bleeding is considered to be high according to clinical evaluation of the ED physician and according to local standard-of-care and clinical practice. The execution of serial CT scans can be time consuming, expensive for the health-care services, and might pose a significant radiological risk for patients; furthermore, this risk might be unjustified considering that the prevalence of development of late intra-cranial bleeding in patients with risk factors who perform a second head CT scan during observation in the ED is considered to be around 2%.

Nonetheless, in this category of patients, clinical observation and the repetition of a second head CT scan is felt to be the safest course of action for patients in order not to overlook potentially fatal injuries.

Ideally, a clinical decision algorithm which takes into consideration a serum biomarker with a high negative predictive value for brain injury might aid the clinician to reduce the number of useless CT scans, therefore reducing the observation time in the ED as well as the exposure to ionizing radiations for the patients, while not increasing the number of missed delayed bleedings.

At present, the role of GFAP and UCH-L1 in the risk stratification of patients with risk factors for delayed cerebral bleeding after mTBI has not been evaluated yet.

DETAILED DESCRIPTION:
Study design Ambispective observational study without drug nor device.

Population The study population will include all non-pregnant patients, who are > 18 y.o. and meet the pre-specified inclusion criteria. We will enroll patients who present to our ED with mTBI and who undergo a venous blood sample and serial brain CT scans as part of their standard emergency care according to the present intra-hospital guidelines and the choice of the attending physician.

Study duration The duration of the study will be of 18 months starting from the approval of the present protocol by the local Ethics Committee of Fondazione Policlinico Universitario Agostino Gemelli IRCCS of Rome. Retrospectively enrolled patients will cover the period from October 2022 up to approval of the protocol, date in which the prospective enrollment will start. The enrolment phase will last 12 months, whilst the following 6 will be dedicated to data extraction, statistical analysis and scientific reporting.

Variables and procedures Retrospective data will be retrieved from our healthcare electronic system for all patients who presented to the ED with the inclusion criteria. In this case, patients will be contacted by phone to provide informed consent. Prospectively enrolled patients will be selected by the attending physician at the moment of the first visit if eligible and written informed consent will be obtained. Patients will be enrolled if they undergo serial CT scans during the emergency evaluation as part of the standard ED care and if a sample of venous blood will be obtained at the moment of the visit. Serum analysis will be performed and dosage of GFAP and UCH-L1 obtained.

The collected variables will cover the following data:

* Demographic and anamnestic data (age, gender, BMI, past comorbidities, etc…);
* Description of the traumatic event and the time elapsed from the event to the first medical evaluation and blood sample;
* Clinical presentation at the moment of the first medical evaluation (including vital parameters and Glasgow Coma Scale);
* Result of the head CT scans performed during the ED visit, as well as the time at which they are performed. The result will be considered as a categorical variable, positive vs negative CT scan, where positive will considered any detected traumatic anomaly regardless of the severity of the injury;
* Serum dosage of GFAP and UCH-L1 obtained at the moment of the visit;
* Duration of ED visit;

Complications during the ED stay:

* Neurological deterioration, defined as a decrease in GCS with respect to the arrival;
* Need for neurosurgical consultation;
* Development of seizures;
* Emergent neurosurgical intervention: craniotomy, hematoma evacuation, need for invasive intra-cranial pressure monitoring, etc…
* Need for emergent airway management due to coma;
* Need for ICU admission;
* Death for any reason.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old;
* Patients who present to the ED within 4 hours since a traumatic event and reporting mTBI.
* Patients who own risk factors for delayed intracranial bleeding, defined as: history of anticoagulant therapy (VKA or DOACs) or known coagulopathy.
* Patients who undergo serial CT scan during the emergency evaluation as part of the standard ED care and if a sample of venous blood will be obtained at the moment of the visit.
* Signed written informed consent to study participation and personal data treatment.

Exclusion Criteria:

* Age <18 years old;
* Pregnant women;
* Refusal to sign written informed consent to study participation and personal data treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all non-pregnant patients, who are > 18 y.o. and meet the pre-specified inclusion criteria. We will enroll patients who present to our ED with mTBI and who undergo a venous blood sample and serial brain CT scans as part of their standard emergency care according to the present intra-hospital guidelines and the choice of the attending physician
Sampling Method: Non-Probability Sample
Enrollment: 1510 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Biomarkers | 30 days
  Sensitivity of the two pre-specified serum biomarkers for the detection of CT scan abnormalities in patients who present to the ED with mTBI and risk factors for delayed bleeding.

SECONDARY OUTCOMES:
Negative predictive value of Biomarkers | 30 days
  Negative predictive value of the two pre-specified serum biomarkers for the detection of CT scan abnormalities in patients who present to the ED with mTBI and risk factors for delayed bleeding
Correlation of biomarkers with composite clinical outcome | 30 days
  • To evaluate the correlation of serum biomarkers with the composite outcome of patients (i.e. composite of neurosurgical consultation, neurological deterioration defined as decrease of GCS during ED observation, development of epileptic seizures, need for neurosurgical intervention (including craniotomy, hematoma evacuation, need for invasive monitoring of intra-cranial pressure), need of airway management and/or ICU admission, death for any reason), as well as single components

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spaziani G, Rozzi G, Baroni S, Napoli G, De Ninno G, Polla DD, Bonadia N, De Matteis G, Piccioni A, Pepa GMD, Urbani A, Gasbarrini A, Franceschi F, Covino M. Prognostic value of GFAP and UCHL-1 biomarkers in high-risk mild traumatic brain injury: A prospective longitudinal study of short- and long-term outcomes. Am J Emerg Med. 2025 Dec 22;101:41-47. doi: 10.1016/j.ajem.2025.12.021. Online ahead of print. PMID 41455435